CLINICAL TRIAL: NCT01835483
Title: A Multicenter Clinical Study to Determine the Performance Characteristics of the MassPLEX Factor II and Factor V Leiden Genotyping Test in Patients With Suspected Thrombophilia
Brief Title: Determination of Performance Characteristics of the MassPLEX Factor II/V Leiden Test
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM-FVL-300
Record Dates: First submitted 2013-04-10; First posted 2013-04-19 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Factor V Leiden; Factor II; Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — De-identified banked genomic DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
To establish the overall agreement of the MassPLEX Factor II and Factor V Leiden Genotyping Test with bi-directional DNA sequencing for Factor II and Factor V Leiden.

DETAILED DESCRIPTION:
De-identified banked genomic DNA samples derived from whole blood from subjects with suspected thrombophilia will be collected from one or more clinical sites. Three clinical laboratory sites will analyze the samples with the FII/FVL Test. Bi-directional DNA sequencing will be performed on all samples at an independent core reference laboratory.

ELIGIBILITY:
Inclusion Criteria:

* suspected thrombophilia
* 18 years of age or older

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected thrombophilia
Sampling Method: Probability Sample
Enrollment: 867 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Performance of the MassPLEX Factor II/V Leiden Test | Samples are collected at time of suspected thrombotic event.
  Overall percent agreement of the FII/FVL Test results to the bi-directional DNA sequencing results.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Sequenom Center for Molecular Medicine, Grand Rapids, Michigan
  - Oregon Health & Science University, Portland, Oregon
  - The Methodist Hospital Research Institute, Houston, Texas